CLINICAL TRIAL: NCT03957356
Title: Single Center, Single Arm, Open-label, Exploratory Clinical Trial to Evaluate the Safety and Efficacy of HLBLS-200 in Patients Requiring Hemostatic Technique for Oozing Hemorrhage During Liver Resection
Brief Title: Study to Evaluate the Safety and Efficacy of HLBLS-200 in Patients Requiring Hemostatic Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HLB Cell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LL-MD-01
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Hemorrhage
Keywords: Hemostatic; Blood oozing; Absorbent hemostatic; Liver resection; Intraperitoneal surgery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Single Arm, Open Label, Single Center Exploratory Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLBLS-200 (Experimental): HLBLS-200, absorbent hemostactic powder, will be applied intraoperatively to stop blood oozing during hepatic resection.
  Interventions: Device: HLBLS-200

INTERVENTIONS:
Device: HLBLS-200 — The amount of HLBLS-200 applied will be determined by the investigator based on the resection area.

SUMMARY:
This is a prospective, open-label, exploratory clinical trial designed to investigate the safety and efficacy of HLBLS-200 (an investigational hemostatic agent). The study will recruit approximately 8 subjects.

DETAILED DESCRIPTION:
Patients scheduled for hepatic resection who voluntarily agree to participate the study will be recruited for the screening procedures.

Patients who meet the eligibility criteria will be assigned to the study. Subjects will receive HLBLS-200 as a supplementary hemostatic technique for oozing hemorrhage which can be occurred during hepatic resection.

A dose of HLBLS-200 based on the area of liver resection will be applied and time to hemostasis of blood oozing will be evaluated.

Patients will be followed for 12 weeks after application of HLBLS-200 to monitor any adverse event.

Study objective:

1. To investigate the safety of HLBLS-200 application.
2. To explore hemostatic function of HLBLS-200 in patients receiving hepatectomy.

ELIGIBILITY:
Inclusion Criteria: (during screening period)

* Subject aged between 18 and 80 years old and scheduled for non-emergent hepatic resection.
* Subject is willing to provide written consent and able to comply with study procedures.
* Female subject of childbearing potential who is willing to use an adequate method of contraception or to be abstinent during the course of the study.

Inclusion Criteria: (during hepatectomy)

* Subjects who need to receive additional hemostatic treatment for blood oozing at the resection site after application of primary hemostatic methods.

Exclusion Criteria: (during screening period)

* Subject with a history of bleeding disorder, platelet disorder or bone marrow disorder.
* Platelet count < 50 X 10^9/L or International normalized ratio > 2.
* Subject who received any drug affecting hemorrhage and/or hemostasis such as anticoagulants, antiplatelet agents or thrombolytic agent within 2 weeks prior to hepatectomy.
* Subject with a history of hypersensitivity to the substance of the investigational device.
* Creatinine clearance < 30mL/min
* Aspartate transaminase or alanine aminotransferase ≥ 3.0 X upper limit of normal.
* Subject with a suspected disorder of decrease in fibrinolytic activity such as disseminated intravascular coagulation.
* Subject with a history of alcohol or drug abuse.
* Pregnant or lactating women
* Subject who have participated in other clinical trial and have received investigation drugs or devices within 4 weeks prior to participation in the study.
* Subject who were judged by the investigator as inadequate for participation in the study.

Exclusion Criteria: (during hepatectomy)

* Subject with following major bleeding (e.g. spurting hemorrhage, hemorrhage from hepatic veins) despite application of primary hemostatic methods
* Subject who is deemed to need anticoagulant treatment within 48 hours of hepatectomy.
* For other reason, subject who were judged by the investigator as inadequate for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Hemostasis at the target blood oozing site | within 3 minutes
  Proportion of participants achieving hemostasis within 3 minutes after HLBLS-200 application
Adverse Event | up to 12 weeks
  Incidence of Adverse Event after application of HLBLS-200

SECONDARY OUTCOMES:
Hemostasis at the target blood oozing site | within 10 minutes
  Proportion of participants achieving hemostasis within 5, 7, 10 minutes after HLBLS-200 application
Time to hemostasis | within 10 minutes
  Time to hemostasis at the target blood oozing site after HLBLS-200 application
Proportion of participants with abnormal laboratory value | up to 12 weeks
  Safety evaluation
Proportion of participants with operation site bleeding after hepatectomy | up to 12 weeks
  Hemorrhage at the operation site

CONTACTS AND LOCATIONS:
Overall Officials: Dongho Choi, MD, Ph.D, Principal Investigator — Hanyang Univ. Medical Center
Locations (1):
- Hanyang Univ. Medical Center, Seoul, South Korea